CLINICAL TRIAL: NCT05500755
Title: Clinical and Radiographic Evaluation of Dentsply Sirona PrimeTaper Implants: A Prospective Medium Term Study
Brief Title: Clinical and Radiographic Evaluation of Dentsply Sirona PrimeTaper Implants
Status: Recruiting | Type: Observational
Sponsor: Aula Dental Avanzada (Other)
Responsible Party: Principal Investigator, Guillem Esteve-Pardo, Principal Investigator, Aula Dental Avanzada
Other Study IDs: DSPT
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Dental Implants
Keywords: Dental implant; Complication; DS Prime Taper

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients DS Prime Taper: Patients who receive al least one DS Prime Taper on his dental implant treatment.
  Interventions: Device: Implant Treatment

INTERVENTIONS:
Device: Implant Treatment — Surgical placement of a DS Prime Taper implant and its posterior prosthesis.
  Other Names: Implant surgery; Implant prosthesis; Implant placement

SUMMARY:
The DS Prime Taper EV dental implant system was recently launched on the implant market by Dentsply Sirona (York, PA, USA).

Dental implant systems are undergoing rapid evolution, ultimately driven by their broad therapeutic indications. As manufacturers strive to keep up with the demands of a growing market, designs are changing faster than clinical evaluation. This means that the time needed to assess medium- and long-term clinical outcomes before designs change again cannot be met.

Clinicians need to have a "real" analysis of the clinical performance of implants before using them. Therefore, reporting of results is necessary to avoid use in patients without proper practical checks even before the recommended 10- and 15-year follow-up periods.

DETAILED DESCRIPTION:
The DS PrimeTaper implant has macro-design features that differ from its predecessor, the OsseoSpeed EV implant (AstraTech Implant System EV, Dentsply Implants, Mölndal, Sweden) with which they share a common surface and internal connection.

Its macro-design has been modified through the introduction of variable thread forms and a more pronounced taper, ultimately making it more aggressive in terms of cutting ability.

While its predecessor, the OsseoSpeed EV implant, has sufficient scientific support, this new system recently introduced on the market does not. All the scientific contributions that can be made will therefore be a first guide for the clinician who wishes to start using this dental implant system.

ELIGIBILITY:
Inclusion Criteria:

* All the patients whom received at least one DS Prime Taper implant.

Exclusion Criteria:

* When dental implant surgery is contraindicated.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients receiving DS Prime Taper dental implant in a private dental office.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Implant Survival Rate | through study completion, an average of 1 year
  Time of survival of DS Prime Taper dental implant placed
Implant Success Rate | through study completion, an average of 1 year
  Radiological assessment of Marginal Bone Levels around DS Prime Taper implants in function
Biological and mechanical complications events | through study completion, an average of 1 year
  All type of complications that may occur during implant survival

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Esteve-Pardo, PhD, Principal Investigator — Clínica Dental Esteve
Locations (1):
- Clínica Dental esteve, Alicante, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available on request from the corresponding author once publication is accomplished.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Once study completion date reached

REFERENCES:
- [Background] Stanford CM, Barwacz C, Raes S, De Bruyn H, Cecchinato D, Bittner N, Brandt J. Multicenter Clinical Randomized Controlled Trial Evaluation of an Implant System Designed for Enhanced Primary Stability. Int J Oral Maxillofac Implants. 2016 Jul-Aug;31(4):906-15. doi: 10.11607/jomi.4869. PMID 27447160
- [Background] Choi NH, Yoon HI, Kim TH, Park EJ. Improvement in Fatigue Behavior of Dental Implant Fixtures by Changing Internal Connection Design: An In Vitro Pilot Study. Materials (Basel). 2019 Oct 7;12(19):3264. doi: 10.3390/ma12193264. PMID 31591290
- [Background] Toia M, Galli S, Cecchinato D, Wennerberg A, Jimbo R. Clinical Evidence of OsseoSpeed EV Implants: A Retrospective Study and Characterization of the Newly Introduced System. Int J Periodontics Restorative Dent. 2019 November/December;39(6):863-874. doi: 10.11607/prd.2549. Epub 2017 Aug 23. PMID 28834532